CLINICAL TRIAL: NCT05303961
Title: A Dose-block Randomized, Double-blind, Placebo/Active-controlled, Single/Multiple Dosing, Dose-escalation Phase I Clinical Trial to Investigate the Safety/Tolerability and Pharmacokinetics of SA001 After Oral Administration in Healthy Male Subjects
Brief Title: Clinical Study to Investigate the Pharmacokinetics and Safety/Tolerability of SA001 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samjin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SJSA001_02
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Healthy
MeSH Terms: interventions — rebamipide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SA001 (Experimental): Part 1: 24 subjects are assigned to single dose groups(240mg, 480mg, 720mg, 1080mg of SA001) in a ratio of 1:1:1:1 and receiving each dose of SA001 in the period 1.
  Part2: 18 subjects are assinged to multiple dose groups(360mg, 720mg, 1080mg of SA001) in a ratio of 1:1:1 and receiving each dose of SA001.
  Interventions: Drug: SA001 240mg + Rebamipide 200mg or Placebo; Drug: SA001 480mg or Placebo; Drug: SA001 710mg + Rebamipide 600mg or Placebo; Drug: SA001 1,080mg or Placebo; Drug: SA001 360mg or Placebo; Drug: SA001 720mg or Placebo
- Rebamipide (Active Comparator): Part 1: 12 subjects are assigned to single dose groups(200mg, 600mg of Rebamipide) in a ratio of 1:1 and receiving each dose of Rebamipide in the period 2.
  Interventions: Drug: SA001 240mg + Rebamipide 200mg or Placebo; Drug: SA001 710mg + Rebamipide 600mg or Placebo
- Placebo (Placebo Comparator): Part 1: 8 subjects receiving a single dose of Placebo in the period 1.
  Part2: 6 subjects receiving multiple dose of Placebo.
  Interventions: Drug: SA001 240mg + Rebamipide 200mg or Placebo; Drug: SA001 480mg or Placebo; Drug: SA001 710mg + Rebamipide 600mg or Placebo; Drug: SA001 1,080mg or Placebo; Drug: SA001 360mg or Placebo; Drug: SA001 720mg or Placebo

INTERVENTIONS:
Drug: SA001 240mg + Rebamipide 200mg or Placebo — Cohort 1 in the Part1(Single dose): Study drug(SA001 240mg + Rebamipide 200mg), Comparator: Placebo
Drug: SA001 480mg or Placebo — Cohort 2 in the Part1(Single dose): Study drug(SA001 480mg), Comparator(Placebo)
  Arms: Placebo; SA001
Drug: SA001 710mg + Rebamipide 600mg or Placebo — Cohort 3 in the Part1(Single dose): Study drug(SA001 720mg + Rebamipide 600mg), Comparator(Placebo)
Drug: SA001 1,080mg or Placebo — Cohort 4 in the Part1(Single dose): Study drug(SA001 1,080mg), Comparator(Placebo)
  Arms: Placebo; SA001
Drug: SA001 360mg or Placebo — Cohort 5 in the Part2(Multiple dose): Study drug(SA001 360mg), Comparator(Placebo)
  Arms: Placebo; SA001
Drug: SA001 720mg or Placebo — Cohort 6 in the Part2(Multiple dose): Study drug(SA001 720mg), Comparator(Placebo)
  Arms: Placebo; SA001
Drug: SA001 1,080mg or Placebo — Cohort 7 in the Part2(Multiple dose): Study drug(SA001 1,080mg), Comparator(Placebo)
  Arms: Placebo; SA001

SUMMARY:
This study consists of Part 1 followed Part 2.

Part 1 The purpose of this phase1 study is to investigate the pharmacokinetics, safety and tolerability of a single oral dose of SA001 and active comparator(Rebamipide) in healthy male volunteers.

Part 2 The purpose of this phase1 study is to investigate the pharmacokinetics, safety and tolerability of multiple oral dose of SA001 in healthy male volunteers.

DETAILED DESCRIPTION:
Part 1(Single dose, dose escalation study, SA001 240mg~1,080mg dose group)

The starting dose is SA001 240mg, and the maximum dose is 1,080mg. Each dose group is assigned to Experimental group (SA001 or SA001 + Active Comparator(Rebamipide)) or Placebo group in a ratio of 3:1. The pharmacokinetics, safety and tolerability of SA001 and its metabolite are investigated after a single oral administration.

Part 2 (Multiple dose, dose escalation study, SA001 360mg~1,080mg dose group)

The starting dose is SA001 360mg, and the maximum dose is 1,080mg. Each dose group is assigned to SA001 or Placebo in a ratio of 3:1. The pharmacokinetics, safety and tolerability of SA001 and its metabolite are investigated after a multiple oral administration.

ELIGIBILITY:
Inclusion Criteria:

1. 19 years to 45 years (Healthy male Korean)
2. Body weight of 55 to 90kg; and BMI of 18.0 to 27.0 kg/m2
3. Subject who voluntarily agrees to participate in this study and has given a written informed consent, after fully understanding the detailed explanation of this study

Exclusion Criteria:

1. Subject with a disease history of any clinically significant condition as below.

   - Liver, Kidney, nervous system, immune system, respiratory system, endocrine system, tumor, cardiovascular disease or mental illness (mood disorder or obsessive-compulsive disorder etc.) etc.
2. Subject with a history of gastrointestinal disease (Crohn's disease, ulcer, acute or chronic pancreatitis, etc.) or gastrointestinal surgery (except simple appendicectomy or hernia surgery) that may affect the absorption of the study drug
3. Subject with a history of clinically significant hypersensitivity or hypersensitivity reactions to drugs (aspirin, antibiotics, etc.)
4. Serum ALT(SGPT)/AST(SGOT) >1.5×institutional upper limit normal (ULN)
5. eGFR< 90mL/min/1.73m2
6. Systolic blood pressure <100 mmHg or >160 mmHg
7. Diastolic blood pressure <60 mmHg or >100 mmHg
8. Inadequate cardiac function confirmed by 12-lead ECG findings at screening as followings:

   * QTcF > 430msec (males)
   * PR interval > 200msec or < 110msec
   * QRS complex > 120msec
   * Evidence of 2nd- or 3rd-degree atrioventricular (AV) block
   * Pathologic Q waves (defined as Q-wave > 40msec or depth > 0.5mV)
   * Evidence of ventricular preexicitation, left bundle branch block (LBBB), right bundle branch block (RBBB, Incomplete RBBB)
9. Subject with risk factors for Torsade de pointes such as long QT syndrome, family history of sudden death, heart failure, hypokalemia, and arrhythmias
10. Subject with a history of drug abuse within 60 days prior to screening or who is positive for drugs of abuse in urine tests at screening
11. Subject who received any drugs such as

    * Prescription drug or herbal medicine within 14 days prior to the first administration of the investigational products
    * Over the counter (OTC) or vitamin within 7 days prior to the first administration of the investigational products
12. Subject who received other investigational products within 90 days prior to the first administration of the investigational products
13. Subject who have donated whole blood within 60 days prior to the first administration of the investigational products, or donated component blood or have received blood transfusion within 30 days prior to the first administration of the investigational products
14. Subject who continuously drink alcohol (more than 21 units/week, 1 unit = 10 g of pure alcohol) or cannot abstain from alcohol during the study period
15. Subject with history of smoking within 90 days prior to the first administration of the investigational products
16. Subject who cannot prohibit grapefruit/ caffeine-containing foods during the study period from 3 days before the first administration of the investigational products
17. Man of reproductive potential not willing to use contraceptive measures during the study period
18. Subject not eligible for study participation in the opinion of the investigator

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2016-06-07 (Actual); Primary Completion 2016-11-11 (Actual); Study Completion 2016-11-11 (Actual)

PRIMARY OUTCOMES:
Measure the Area Under the plasma concentration versus time Curve from the first observed to last(AUClast) of SA001 and Rebamipide | Part 1: Predose(Day 1 0hour, Day 15 0hour), Postdose(Day 1 0.25~48hours, Day 15 0.25~48hours)
  Investigate the pharmacokinetic parameters by collecting blood before and during administration of the investigational product.
Measure the Area Under the plasma concentration versus time Curve from the first sampled data extrapolated to infinity(AUCinf) of SA001 and Rebamipide | Part 1: Predose9Day 1 0hour, Day 15 0hour), Postdose(Day 1 0.25~48hours, Day 15 0.25~48hours)
  Investigate the pharmacokinetic parameters by collecting blood before and during administration of the investigational product.
Measure the Peak Plasma Concentration (Cmax) of SA001 and Rebamipide | Part 1: Predose(Day 1 0hour, Day 15 0hour), Postdose(Day 1 0.25~48hours, Day 15 0.25~48hours)
  Investigate the pharmacokinetic parameters by collecting blood before and during administration of the investigational product.
Measure the Time to peak drug concentration(Tmax) of SA001 and Rebamipide | Part 1: Predose(Day 1 0hour, Day 15 0hour), Postdose(Day 1 0.25~48hours, Day 15 0.25~48hours)
  Investigate the pharmacokinetic parameters by collecting blood and urine before and during administration of the investigational product.
Measure the Half Life(t1/2) of SA001 and Rebamipide | Part 1: Predose(Day 1 0hour, Day 15 0hour), Postdose(Day 1 0.25~48hours, Day 15 0.25~48hours)
  Investigate the pharmacokinetic parameters by collecting blood before and during administration of the investigational product.
Measure the apparent total body clearance(CL/F) of SA001 and Rebamipide | Part 1: Predose(Day 1 0hour, Day 15 0hour), Postdose(Day 1 0~48hours, Day 15 0~24hours)
  Investigate the pharmacokinetic parameters by collecting urine before and during administration of the investigational product.
Measure the apparent volume of distribution(Vz/F) of SA001 and Rebamipide | Part 1: Predose(Day 1 0hour, Day 15 0hour), Postdose(Day 1 0~48hours, Day 15 0~24hours)
  Investigate the pharmacokinetic parameters by collecting urine before and during administration of the investigational product.
Measure the Renal Clearance(CLr) of SA001 and Rebamipide | Part 1: Predose(Day 1 0hour, Day 15 0hour), Postdose(Day 1 0~48hours, Day 15 0~24hours)
  Investigate the pharmacokinetic parameters by collecting urine before and during administration of the investigational product.
Measure the cumulative fraction excreted unchanged parent in urine(Fe) of SA001 and Rebamipide | Part 1: Predose(Day 1 0hour, Day 15 0hour), Postdose(Day 1 0~48hours, Day 15 0~24hours)
  Investigate the pharmacokinetic parameters by collecting urine before and during administration of the investigational product.
Measure the Trough Drug Concentration at steady state(Cmin,ss) of SA001 | Part 2: Predose(Day 1 0, 12hour, Day 2 0hour, Day 5 0hour, Day 7 12hour, Day 8 0, 12hour), Postdose(Day 1 0.25~8hours, Day 8 0.25~8hours)
  Investigate the pharmacokinetic parameters by collecting blood before and during administration of the investigational product.
Measure the Peak Plasma Concentration at steady state(Cmax,ss) of SA001 | Part 2: Predose(Day 1 0, 12hour, Day 2 0hour, Day 5 0hour, Day 7 12hour, Day 8 0, 12hour), Postdose(Day 1 0.25~8hours, Day 8 0.25~8hours)
  Investigate the pharmacokinetic parameters by collecting blood before and during administration of the investigational product.
Measure the average drug concentration in plasma during a dosing interval at steady state(Cav,ss) of SA001 | Part 2: Predose(Day 1 0, 12hour, Day 2 0hour, Day 5 0hour, Day 7 12hour, Day 8 0, 12hour), Postdose(Day 1 0.25~8hours, Day 8 0.25~8hours)
  Investigate the pharmacokinetic parameters by collecting blood before and during administration of the investigational product.
Measure the area under the plasma concentration-time curve for dosing interval(AUCτ) of SA001 | Part 2: Predose(Day 1 0, 12hour, Day 2 0hour, Day 5 0hour, Day 7 12hour, Day 8 0, 12hour), Postdose(Day 1 0.25~8hours, Day 8 0.25~8hours)
  Investigate the pharmacokinetic parameters by collecting blood before and during administration of the investigational product.
Measure the Time to peak drug concentration at steady state(Tmax,ss) of SA001 | Part 2: Predose(Day 1 0, 12hour, Day 2 0hour, Day 5 0hour, Day 7 12hour, Day 8 0, 12hour), Postdose(Day 1 0.25~8hours, Day 8 0.25~8hours)
  Investigate the pharmacokinetic parameters by collecting blood before and during administration of the investigational product.
Measure the Half Life(t1/2) of SA001 | Part 2: Predose(Day 1 0, 12hour, Day 2 0hour, Day 5 0hour, Day 7 12hour, Day 8 0, 12hour), Postdose(Day 1 0.25~8hours, Day 8 0.25~8hours)
  Investigate the pharmacokinetic parameters by collecting blood before and during administration of the investigational product.
Measure the Peak-trough Fluctuation (PTF) of SA001 | Part 2: Predose(Day 1 0, 12hour, Day 2 0hour, Day 5 0hour, Day 7 12hour, Day 8 0, 12hour), Postdose(Day 1 0.25~8hours, Day 8 0.25~8hours)
  Investigate the pharmacokinetic parameters by collecting blood before and during administration of the investigational product.
Measure the Fraction recovered unchanged in urine (FR) of SA001 | Part 2: Predose(Day 1 0hour, Day 8 0hour, Day 16 0hour), Postdose(Day 1 0~24hours, Day 8 0~24hours, Day 16 0~24hours, Day 17 0~24hours)
  Investigate the pharmacokinetic parameters by collecting urine before and during administration of the investigational product.
Measure the apparent total body clearance(CL/F) of SA001 | Part 2: Predose(Day 1 0hour, Day 8 0hour, Day 16 0hour), Postdose(Day 1 0~24hours, Day 8 0~24hours, Day 16 0~24hours, Day 17 0~24hours)
  Investigate the pharmacokinetic parameters by collecting urine before and during administration of the investigational product.
Measure the Renal Clearance(CLr) of SA001 | Part 2: Predose(Day 1 0hour, Day 8 0hour, Day 16 0hour), Postdose(Day 1 0~24hours, Day 8 0~24hours, Day 16 0~24hours, Day 17 0~24hours)
  Investigate the pharmacokinetic parameters by collecting urine before and during administration of the investigational product.

SECONDARY OUTCOMES:
Incidence of Adverse Event(AE) | Part 1: Day-1(before the administration) to approximately Day 24 (Post study Visit) / Part 2: Day-1(before the administration) to approximately Day 29 (Post study Visit)
  Safety/Tolerability Assessment